CLINICAL TRIAL: NCT02532985
Title: A Randomized, Double-Blind, Crossover Study to Assess Gastrointestinal Tolerability of Cba-1, a Novel Dietary Fiber, Using Three Dose Levels at Multiple Eating Occasions in Healthy Men and Women
Brief Title: Gastrointestinal Tolerability Following Multiple Servings of a Novel Dietary Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: BIO-1411
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Gastrointestinal tolerability; dietary fiber; clinical trial; healthy subjects
MeSH Terms: conditions — Signs and Symptoms, Digestive | interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Negative control (Placebo Comparator): No added fiber
  Interventions: Other: Negative Control
- Positive fiber control (Active Comparator): 90g positive control fiber
  Interventions: Other: Positive Fiber Control
- Novel fiber 30g (Experimental): 30g novel fiber
  Interventions: Other: Novel Fiber
- Novel fiber 60g (Experimental): 60g novel fiber
  Interventions: Other: Novel Fiber
- Novel fiber 90g (Experimental): 90g novel fiber
  Interventions: Other: Novel Fiber

INTERVENTIONS:
Other: Negative Control — No added fiber beverage
  Arms: Negative control
Other: Positive Fiber Control — positive control fiber supplemented beverage provided over 4 servings
  Other Names: Polydextrose
  Arms: Positive fiber control
Other: Novel Fiber — novel fiber supplemented beverage provided over 4 servings
  Other Names: Cba-1
  Arms: Novel fiber 30g
Other: Novel Fiber — novel fiber supplemented beverage provided over 4 servings
  Other Names: Cba-1
  Arms: Novel fiber 60g
Other: Novel Fiber — novel fiber supplemented beverage provided over 4 servings
  Other Names: Cba-1
  Arms: Novel fiber 90g

SUMMARY:
The study will assess the gastrointestinal tolerability of multiple servings of a novel dietary fiber at three different dose levels in generally healthy men and women. Double-blind controlled, cross-over clinical trial with negative (no added fiber) and positive controls. Multiple servings over 24h, with data collection at 24 and 48h and 1 week wash-out between cross-overs. 45 randomized, generally healthy men and women, 18-54 y, BMI higher or equal to 18.5 and smaller or equal to 39.99 kg/m2. Novel dietary fiber ingredient and positive control will be delivered in 240 ml beverages.

DETAILED DESCRIPTION:
This is a randomized, double-blind, five test periods crossover study consisting of a screening visit (visit 1, day -7) and 10 test visits (days 0, 2, 7, 9, 14, 16, 21, 23, 28, 30). At the screening visit, after subjects have provided informed consent, medical history and clinic visit procedures will be performed. Subjects who meet the study criteria will be instructed to maintain habitual diet and physical activity patterns throughout the study period. Subjects will also be instructed to avoid foods/ beverages that cause Gastrointestinal (GI)-distress, as well as high-fiber foods for the 24 h prior to and throughout each 48 h test period. Additional instructions will include avoiding the use of non-steroidal anti-inflammatory drugs (NSAIDS), antacids, proton pump inhibitors (PPIs), and H2 receptor antagonists for the 48 h prior to the next clinic visit (visit 2, day 0). At the test visits, eligible subjects will undergo clinic visit procedures, including assessment of adverse events (AEs).

At the beginning of each test period (Visits 2, 4, 6, 8, and 10), subjects will arrive at the clinic after a 9-14 h fast and will be administered one serving of their assigned study product to consume within 15 min with a standard breakfast meal (t = 0 h). Subjects will remain in the clinic and will be provided a second serving of their assigned study product to consume within 15 min with a standard lunch meal at t= 4 ± 0.5 h. Subjects will then be provided the third and fourth servings of their assigned study product and instructed to consume the study product in its entirety within 15 min of their also provided afternoon snack, and evening dinner, respectively, and to allow at least 3 h between eating occasions. Compliance with dispensed product and meal consumption will be confirmed with a diet record. Subjects will be also instructed to complete a GI Tolerability Questionnaire the next morning (t=24h) after an overnight fast (9-14h). A Bowel Habits Diary will be completed from the initial study product consumption (t= 0) until the subsequent clinic visit (t= 48 h). Subjects will return to the clinic at t= 48 h (Visits 3, 5, 7, 9, and 11) after an overnight fast (9-14 h) to complete the test period, at which time a 48 h GI Tolerability Questionnaire will also be completed.

A washout period of 7 d will occur between each test period (e.g., before Visits 4, 6, 8, and 10), after which subjects will return to the clinic to cross over to the next study product in their test sequence.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18-54 years of age, inclusive.
* Subject has body mass index (BMI) ≥18.50 and ≤39.99 kg/m2 at visit 1 (day -7) and has been weight stable (± 4.5 kg) for the previous 3 months.
* Subject is judged to be in good health on the basis of medical history.
* Subject is willing to maintain his or her habitual diet and physical activity patterns, including habitual use of study approved medications and/or dietary supplements throughout the study period.
* Subject is willing to avoid foods/beverages that cause GI-distress, as well as high-fiber foods for 24 h prior to test visits.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

* Subject reports any clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, history of surgery for weight loss, gastroparesis, and clinically important lactose intolerance).
* History or presence of clinically important endocrine (including type 1 or 2 diabetes mellitus), cardiovascular, pulmonary, biliary, renal, hepatic, pancreatic, or neurologic disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* Recent history (within 6 weeks of screening, visit 1) of constipation (defined as <3 bowel movements per week), and/or diarrhea (defined as ≥3 loose or liquid stools/d).
* Recent (within 6 weeks of screening, visit 1) episode of acute GI illness such as nausea, vomiting or diarrhea.
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDS),
* Daily use of antacids, proton pump inhibitors, and/or H2 blockers.
* Recent use of antibiotics (within 3 months of visit 2, day 0).
* Use of medications (over-the-counter and prescription) or dietary supplements (within 3 weeks of visit 2, day 0) known to influence GI function such as constipation medications and supplements (including laxatives, enemas, fiber supplements and/or suppositories); anti-diarrheal agents; anti-spasmodic; prebiotic and probiotic supplements.
* Extreme dietary habits, including but not limited to vegetarian diets and intentional consumption of a high fiber diet.
* Known allergy or sensitivity to food ingredients such as: soy, dairy (milk), wheat, egg, peanuts, tree nuts, fin fish and crustacean.
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg at visit 1, day -7).
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Any major trauma or surgical event within 2 months of visit 2, day 0.
* Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who were unwilling to commit to use of a medically approved form of contraception throughout the study period.
* Exposure to any non-registered drug product within 30 days previous to the screening visit.
* Recent history of (within 12 months of visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Recent history of (within 2 months of visit 1) use of any tobacco-containing products.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Composite Gastrointestinal GI Symptom Score among conditions | 24 hours
  Composite score will be calculated for each intake level as the sum of the ratings of the individual components (abdominal distention/bloating, gas/flatulence, borborygmus/stomach rumbling, and abdominal cramping). The ratings will be coded using a 4-point scale, in which 1 = none, 2 = mild, 3 = moderate, and 4 = severe.
Composite Gastrointestinal GI Symptom Score among conditions | 48 hours
  Composite score will be calculated for each intake level as the sum of the ratings of the individual components (abdominal distention/bloating, gas/flatulence, borborygmus/stomach rumbling, and abdominal cramping). The ratings will be coded using a 4-point scale, in which 1 = none, 2 = mild, 3 = moderate, and 4 = severe.